CLINICAL TRIAL: NCT00429793
Title: A Phase II Evaluation of CCI-779 (Temsirolimus, NCI-Supplied Agent, NSC #683864, IND #61010) in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: Temsirolimus in Treating Patients With Refractory or Recurrent Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02707; NCI-2012-02707 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000528257; GOG-0170I (Other: Gynecologic Oncology Group); GOG-0170I (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Fallopian Tube Cancer; Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temsirolimus

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
This phase II trial is studying the side effects and how well temsirolimus works in treating patients with refractory or recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine the 6-month progression-free survival (PFS) or objective tumor response in patients with refractory or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer treated with temsirolimus.

II. Determine the toxicity of this drug in these patients.

Secondary I. Determine the duration of PFS and overall survival of these patients.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 52 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial, fallopian tube or primary peritoneal cavity cancer

  * Recurrent or refractory
* Prior treatment with ≥ 1 platinum-based chemotherapeutic regimen for management of primary disease (containing carboplatin, cisplatin, or another organoplatinum compound) required

  * Initial treatment may have included any of the following:

    * High-dose therapy
    * Intraperitoneal therapy
    * Consolidation therapy
    * Noncytotoxic agents
    * Extended therapy administered after surgical or nonsurgical assessment
  * Patients must meet ≥ 1 of the following criteria:

    * Treatment-free interval after platinum therapy of < 12 months for patients who received only 1 platinum-based regimen
    * Progressed during platinum-based therapy
    * Refractory disease after a platinum-based regimen
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * Must have ≥ 1 target lesion

    * Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained ≥ 90 days after completion of radiotherapy
* Not eligible for a higher priority GOG protocol, if one exists
* GOG performance status (PS) 0-2 for patients who have receive one prior regimen OR GOG PS 0-1 for patients who have received 2-3 prior regimens
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* No neuropathy (sensory and motor) > grade 2
* Fasting cholesterol < 350 mg/dL
* Fasting triglycerides < 400 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics (with the exception of uncomplicated UTI)
* No other invasive malignancies within the past 5 years, except for non-melanoma skin cancer, breast cancer, or head and neck cancer
* See Disease Characteristics
* Recovered from prior surgery, radiotherapy, or chemotherapy
* At least 1 week since prior hormonal therapy directed at the malignant tumor
* At least 3 years since prior radiotherapy for localized cancer of the breast, head and neck, or skin

  * Patient must remain free of recurrent or metastatic disease
* At least 3 years since prior adjuvant chemotherapy for localized breast cancer

  * Patient must remain free of recurrent or metastatic disease
* At least 3 weeks since other prior therapy directed at the malignant tumor, including immunologic agents
* No prior temsirolimus
* No prior cancer treatment that would preclude study therapy
* No prior radiotherapy to > 25% of marrow-bearing areas
* No prior radiotherapy to any portion of the abdominal cavity or pelvis, except for the treatment of ovarian cancer
* No prior non-cytotoxic therapy for management of recurrent or persistent ovarian disease, except for therapy that was part of the primary treatment regimen
* Two additional cytotoxic regimens (defined as any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa) for management of recurrent or persistent ovarian disease allowed
* Concurrent low molecular weight heparin allowed provided PT/INR ≤ 1.5
* Concurrent hormone replacement therapy allowed
* No concurrent amifostine or other protective reagents
* No concurrent prophylactic filgrastim (G-CSF)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian Behbakht, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Behbakht K, Sill MW, Darcy KM, Rubin SC, Mannel RS, Waggoner S, Schilder RJ, Cai KQ, Godwin AK, Alpaugh RK. Phase II trial of the mTOR inhibitor, temsirolimus and evaluation of circulating tumor cells and tumor biomarkers in persistent and recurrent epithelial ovarian and primary peritoneal malignancies: a Gynecologic Oncology Group study. Gynecol Oncol. 2011 Oct;123(1):19-26. doi: 10.1016/j.ygyno.2011.06.022. Epub 2011 Jul 12. PMID 21752435
- [Derived] Yap TA, Carden CP, Kaye SB. Beyond chemotherapy: targeted therapies in ovarian cancer. Nat Rev Cancer. 2009 Mar;9(3):167-81. doi: 10.1038/nrc2583. PMID 19238149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued to the first stage of accrual from 2/5/07 to 9/4/07. Patients were accrued to the second stage of accrual between 5/7/08 to 8/25/08. They received 25 mg IV of CCI-779 weekly. One cycle was 28 days.
Pre-assignment Details: Patients were required to have had one regimen of a platinum agent for the treatment of ovarian cancer. Patients entering the study therefore were required to have either persistent or recurrent cancer that was measurable by RECIST.
Period: Overall Study
Arm/Group | Treatment (Temsirolimus)
Started | 60
Completed | 54
Not Completed | 6
Not completed — Improper pre-protocol treatment | 3
Not completed — Required test not done | 1
Not completed — Never treated | 1
Not completed — Non-measurable | 1

BASELINE CHARACTERISTICS:
Population: Number of eligible and evaluable participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (13.0)
Age, Customized [Number; unit: participants]
  20-29 years | 2
  40-49 years | 7
  50-59 years | 15
  60-69 years | 11
  70-79 years | 16
  80-89 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 54
International Federation of Gynecology and Obstetrics (FIGO) Recurrent/Persistent Disease [Number; unit: participants] | 54
Cell Type [Number; unit: participants]
  Adenocarcinoma, unspecified | 8
  Clear Cell Carcinoma | 3
  Endometrioid Adenocarcinoma | 4
  Serous Adenocarcinoma | 39

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression-free Survival (PFS)
Description: Number of participants who survived progression-free for more than 6 months.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 54
participants | 13

2. Primary Outcome: Objective Tumor Response Based on the Gynecologic Oncology Group (GOG) Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Number of participants who experienced an objective tumor response up to 5 years. Per RECIST version 1.0 criteria: each target lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI, or >= 10 mm when measured by spiral CT. Complete Response is a disappearance of all target and non-target lesions. Partial Response is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions, taking as reference the baseline sum of LD. Increasing Disease is at least a 20% increase in the sum of LD of target lesions, taking as references the smallest sum LD or the appearance of new lesions.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 54
participants
  Partial Response | 5
  Stable Disease | 22
  Increase Disease | 21
  Indeterminate | 6

3. Primary Outcome: Frequency and Severity of Adverse Events as Assessed by the Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE v3.0)
Time Frame: Up to 5 years
Population: Eligible and evaluable patients.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 1 (CTCAE v3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5 (CTCAE v 3.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 1 (CTCAE v3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5 (CTCAE v 3.0)
Number analyzed (Participants) | 54 | 54 | 54 | 54 | 54
Participants
  Leukopenia | 14 | 14 | 0 | 0 | 0
  Thrombocytopenia | 18 | 5 | 0 | 0 | 0
  Neutropenia | 6 | 12 | 1 | 0 | 0
  Anemia | 20 | 19 | 3 | 0 | 0
  Other hematologic | 0 | 2 | 0 | 0 | 0
  Allergy/Immunology | 1 | 0 | 0 | 0 | 0
  Auditory/Ear | 1 | 0 | 0 | 0 | 0
  Cardiac | 3 | 1 | 1 | 0 | 0
  Coagulation | 2 | 1 | 0 | 0 | 0
  Constitutional | 23 | 15 | 4 | 1 | 0
  Dermatologic | 24 | 10 | 1 | 0 | 0
  Nausea | 19 | 2 | 2 | 0 | 0
  Vomiting | 2 | 3 | 1 | 0 | 0
  Gastrointestinal | 16 | 19 | 6 | 0 | 0
  Genitourinary/Renal | 4 | 0 | 1 | 0 | 0
  Hemorrhage | 5 | 0 | 0 | 0 | 0
  Infection | 0 | 5 | 2 | 0 | 0
  Lymphatics | 3 | 1 | 1 | 0 | 0
  Metabolic | 17 | 12 | 8 | 0 | 0
  Musculoskeletal | 2 | 0 | 1 | 0 | 0
  Neurosensory | 6 | 2 | 0 | 0 | 0
  Other Neurological | 5 | 1 | 0 | 0 | 0
  Ocular/Visual | 1 | 0 | 0 | 0 | 0
  Pain | 13 | 7 | 6 | 0 | 0
  Pulmonary | 17 | 5 | 4 | 0 | 0
  Sexual/Reproductive | 1 | 0 | 0 | 0 | 0
  Vascular | 0 | 0 | 0 | 1 | 0

4. Secondary Outcome: Duration of Progression-free Survival
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months up to 5 years
Population: Eligible and evaluable patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 54
months | 3.19 [1.74 to 5.82]

5. Secondary Outcome: Duration of Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and evaluable patients.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 54
months | 11.60 [6.83 to 22.83]

6. Other Pre Specified Outcome: Reason Off Study Therapy
Time Frame: from study entry until end of study treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 54
participants
  Disease Progression | 37
  Refused Further Treatment | 5
  Toxicity as permitted | 8
  Other | 3
  Unspecified | 1

7. Other Pre Specified Outcome: Patient Vital Status
Description: Patients alive or dead after 24 months from time of study entry
Time Frame: Study entry up to 2 years
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 54
participants
  Alive without disease progression | 5
  Alive with disease progression | 19
  Dead from disease | 29
  Dead from neither treatment nor disease | 1

ADVERSE EVENTS:
Time Frame: All Adverse Events(AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment.
Arm/Group | Treatment (Temsirolimus)
Serious Adverse Events (participants affected / at risk) | 5/54
Other Adverse Events (participants affected / at risk) | 44/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temsirolimus) (N=54)
Fatigue (General disorders) | 1
Insomnia (General disorders) | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 5
Dehydration (Gastrointestinal disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Pain: Head/Headache (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Obstruction, Gu - Bladder (Renal and urinary disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temsirolimus) (N=54)
Tinnitus (Ear and labyrinth disorders) | 5
Neutrophils (Blood and lymphatic system disorders) | 19
Platelets (Blood and lymphatic system disorders) | 24
Leukocytes (Blood and lymphatic system disorders) | 28
Hemoglobin (Blood and lymphatic system disorders) | 44
Fibrinogen (Vascular disorders) | 3
Ptt (Vascular disorders) | 3
Fever (General disorders) | 6
Weight Loss (General disorders) | 9
Rigors/Chills (General disorders) | 3
Fatigue (General disorders) | 43
Insomnia (General disorders) | 5
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 9
Acne (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 25
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6
Hot Flashes (Endocrine disorders) | 7
Heartburn (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 4
Taste Alteration (Gastrointestinal disorders) | 5
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 20
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 13
Anorexia (Gastrointestinal disorders) | 22
Dehydration (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 28
Diarrhea (Gastrointestinal disorders) | 24
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 5
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 9
Edema: Limb (Blood and lymphatic system disorders) | 11
Ast (Metabolism and nutrition disorders) | 15
Cholesterol,serum High (Metabolism and nutrition disorders) | 30
Creatinine (Metabolism and nutrition disorders) | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Alt (Metabolism and nutrition disorders) | 5
Alkaline Phosphatase (Metabolism and nutrition disorders) | 10
Bilirubin (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypertriglyceridemia (Metabolism and nutrition disorders) | 28
Hypocalcemia (Metabolism and nutrition disorders) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hypokalemia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Mood Alteration - Depression (Nervous system disorders) | 8
Mood Alteration - Anxiety (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 6
Neuropathy-Sensory (Nervous system disorders) | 22
Blurred Vision (Eye disorders) | 3
Pain - Other (General disorders) | 3
Pain: Chest /Thorax Nos (General disorders) | 4
Pain: Head/Headache (General disorders) | 12
Pain: Extremity-Limb (General disorders) | 7
Pain: Back (General disorders) | 6
Pain: Joint (General disorders) | 4
Pain: Abdominal Pain Nos (General disorders) | 18
Pain: Muscle (General disorders) | 4
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18
Urinary Frequency (Renal and urinary disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less